CLINICAL TRIAL: NCT03608267
Title: A Prospective Study to Evaluate the Safety and Feasibility of an Endoluminal-suturing Device (Endomina TM) as an Aid for Afferent Loop Syndrome
Brief Title: Safety and Feasibility of Endomina, an Candy Cane Syndrome Endoluminal Suturing Device
Acronym: Endomina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRB_201804_011 -- P2018/336
Record Dates: First submitted 2018-06-15; First posted 2018-07-31 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Bariatric Surgery; Complication
Keywords: endoscopy; mini invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — The jejunum between the two loops is sutered with Endomina and cut 15 days later.

SUMMARY:
Surgery is currently the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Lap Band and Sleeve gastrectomy), malabsorptive surgeries (Biliary pancreatic deviation and duodenal switch) or a combination of both (RYGBP).

This latter technique is the most common and most effective surgical procedure performed worldwide and has been processed to be an effective treatment of morbid obesity and its complications, achieving excess weight loss of 65 to 80 %; 1-2 years after surgery (1,2).

Morbidity after RYGB includes the candy cane syndrome or afferent loop syndrome. Candy cane Roux syndrome in patients who have undergone RYGB refers to an excessively long blind afferent Roux limb at the gastrojejunostomy causing postprandial pain often relieved by vomiting. It is believed that the blind afferent limb ("candy cane") acts as an obstructed loop when filled with food (often preferentially), and the distention of the loop causes pain until the food either spills into the Roux limb or is vomited back out (3).

Patients have been reported presenting as early as three months and as late as 11 years after their initial RYGB, typically with symptoms of postprandial epigastric pain, nausea, vomiting, and reflux or food regurgitation (4). The diagnosis is confirmed by upper gastrointestinal contrast studies or endoscopy. On upper gastrointestinal series, the afferent limb fills before contrast spills into the Roux limb. On upper endoscopy, the afferent limb is usually the most direct outlet of the gastrojejunostomy (3).

The treatment is revision bariatric surgery, most commonly laparoscopic resection of the afferent limb, which ranged in length from 3 to 22 cm in one study (mean of 7.6 cm) (3). Symptoms resolve after revision surgery in most patients. Surgeons should minimize the length of the blind afferent loop left at the time of initial RYGB to prevent candy cane Roux syndrome.

Endomina (Endo Tools Therapeutics, Gosselies, Belgium) is a CE marked device that may be attached to an endoscope inside the body and allows remote actuation of the device during a peroral intervention. It offers the possibilities of making transoral full thickness tissue apposition and may allow performing, via a transoral route, large plications with tight serosa to serosa apposition.

DETAILED DESCRIPTION:
Surgery is currently the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Lap Band and Sleeve gastrectomy), malabsorptive surgeries (Biliary pancreatic deviation and duodenal switch) or a combination of both (RYGBP).

This latter technique is the most common and most effective surgical procedure performed worldwide and has been processed to be an effective treatment of morbid obesity and its complications, achieving excess weight loss of 65 to 80 %; 1-2 years after surgery (1,2).

Morbidity after RYGB includes the candy cane syndrome or afferent loop syndrome. Candy cane Roux syndrome in patients who have undergone RYGB refers to an excessively long blind afferent Roux limb at the gastrojejunostomy causing postprandial pain often relieved by vomiting. It is believed that the blind afferent limb ("candy cane") acts as an obstructed loop when filled with food (often preferentially), and the distention of the loop causes pain until the food either spills into the Roux limb or is vomited back out (3).

Patients have been reported presenting as early as three months and as late as 11 years after their initial RYGB, typically with symptoms of postprandial epigastric pain, nausea, vomiting, and reflux or food regurgitation (4). The diagnosis is confirmed by upper gastrointestinal contrast studies or endoscopy. On upper gastrointestinal series, the afferent limb fills before contrast spills into the Roux limb. On upper endoscopy, the afferent limb is usually the most direct outlet of the gastrojejunostomy (3).

The treatment is revision bariatric surgery, most commonly laparoscopic resection of the afferent limb, which ranged in length from 3 to 22 cm in one study (mean of 7.6 cm) (3). Symptoms resolve after revision surgery in most patients. Surgeons should minimize the length of the blind afferent loop left at the time of initial RYGB to prevent candy cane Roux syndrome.

Endomina (Endo Tools Therapeutics, Gosselies, Belgium) is a CE marked device that may be attached to an endoscope inside the body and allows remote actuation of the device during a peroral intervention. It offers the possibilities of making transoral full thickness tissue apposition and may allow performing, via a transoral route, large plications with tight serosa to serosa apposition.

ELIGIBILITY:
Inclusion Criteria:

1. Proven Candy cane syndrome by barium swallow
2. Age between 18-65 years;
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations;
4. Must be able to understand and be willing to provide written informed consent;
5. Must live within 75 km of the treatment site;
6. Had followed the bariatric multidisciplinary workup (blood analyses, dietician, psychologist and doctor appointments).

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders;
2. Severe esophagitis;
3. Gastro-duodenal ulcer;
4. Severe renal, hepatic, pulmonary disease or cancer;
5. GI stenosis or obstruction;
6. Pregnancy, breastfeeding or willing to become pregnant in the coming 18 months;
7. Anticoagulant therapy;
8. Impending gastric surgery 60 days post intervention;
9. Currently participating in other study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Characterisation of safety by measurement of the incidence of all adverse device effects (ADE) | 6 months
  Incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or the device.
  Definitions are combined from EN ISO 14155:2011 and MEDDEV 2.7/3 rev 3 (May 2015).

SECONDARY OUTCOMES:
Efficacy of the device: Dakkak and Bennett dysphagia score | 6 months
  scoring using the Dakkak and Bennett dysphagia score 0 = no dysphagia; 4= aphagia Total scale will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, MD, Principal Investigator — Erasme University Hospital
Locations (2):
- Belgium (2):
  - CUB Hopital erasme, Anderlecht
  - Gastroenterology Department Erasme Hospital, Brussels

IPD SHARING:
Plan to Share IPD: No